CLINICAL TRIAL: NCT07086820
Title: Window Prophylaxis for Mycobacterium Tuberculosis Infection Prevention in Child and Adolescent Household Contacts: a Cluster-Randomized Controlled Trial
Brief Title: Window Prophylaxis for Pediatric Tuberculosis Prevention Trial
Acronym: TB-WIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, María Elvira Balcells, MD, Associate Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 240519001; FONDECYT N° 1250853 (Other Grant/Funding Number: Agencia Nacional de Investigación y Desarrollo de Chile (ANID))
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis Infection; Household Contacts; Children; Adolescent; Tuberculosis Infection, Latent; Tuberculosis
Keywords: Household contacts; Prophylaxis; Tuberculosis infection; Mycobacterium tuberculosis; Children; Adolescent; Randomized clinical trial; Tuberculosis; Cluster-randomized trial
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Isoniazid; Chemoprevention

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, controlled, cluster-randomized, open-label, superiority trial. A total of 360 households (clusters), each with at least one child aged ≥5 to <18 years and recently exposed to a new case of pulmonary tuberculosis within the household, will be randomly assigned in a 1:1 allocation ratio to either the intervention or control arm.
  The intervention consists of a window prophylaxis strategy, while the control involves prophylaxis only for participants with confirmed M. tuberculosis infection.
  To ensure early enrollment, households will be eligible only if the tuberculosis index patient has received no more than 15 daily doses of antituberculous treatment, for both study arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care tuberculosis prophylaxis (Active Comparator): In the Control Arm, only participants with a positive baseline IGRA result will receive tuberculosis preventive treatment (TPT). Therefore, TPT will not be given to participants with a negative baseline IGRA result at enrollment.
  Interventions: Drug: Standard of care tuberculosis prophylaxis with weekly rifapentine and isoniazid for 12 weeks
- Window tuberculosis prophylaxis (Experimental): In the Intervention Arm, all participants will be immediately prescribed tuberculosis preventive treatment (TPT), irrespective of their baseline IGRA result. Therefore, TPT will be given to participants having either positive or negative baseline IGRA results at enrollment.
  Interventions: Drug: Tuberculosis window prophylaxis with weekly rifapentine and isoniazid for 12 weeks

INTERVENTIONS:
Drug: Tuberculosis window prophylaxis with weekly rifapentine and isoniazid for 12 weeks — Weekly isoniazid and rifapentine for 12 weeks (3HP regimen) will be provided to all participants.
  Other Names: Window prophylaxis; Window period tuberculosis prophylaxis; Universal tuberculosis prophylaxis
  Arms: Window tuberculosis prophylaxis
Drug: Standard of care tuberculosis prophylaxis with weekly rifapentine and isoniazid for 12 weeks — Weekly isoniazid and rifapentine for 12 weeks (3HP regimen) will be provided only to participants with a positive IGRA result at baseline.
  Other Names: Tuberculosis prophylaxis; Chemoprophylaxis; Tuberculosis preventive treatment (TPT)
  Arms: Standard of care tuberculosis prophylaxis

SUMMARY:
The goal of this cluster-randomized controlled trial is to evaluate the effectiveness of tuberculosis preventive treatment (TPT) administered during the "window period" to prevent new Mycobacterium tuberculosis infections in children and adolescents.

The main question it aims to answer is:

Can immediate TPT reduce the incidence of IGRA conversions in children and adolescents who are household contacts of a newly diagnosed pulmonary tuberculosis patient?

Researchers will compare the incidence of new tuberculosis infections-measured by IGRA conversion at 12 weeks-between participants who receive immediate TPT while still uninfected (baseline IGRA-negative) and those who receive standard care, in which TPT is not offered to IGRA-negative contacts.

Participants will be:

1. Tested for M. tuberculosis infection using the Interferon-Gamma Release Assay (IGRA), specifically the QuantiFERON-TB Gold Plus, at enrollment and after 12 weeks of follow-up.
2. Take weekly isoniazid and rifapentine for 12 weeks if:

   1. They are assigned to the intervention arm (regardless of baseline IGRA result), or
   2. They are in the control arm and test IGRA-positive at baseline.

Additionally, participants from the control arm who experience an IGRA conversion at 12 weeks (following the primary outcome assessment) will also receive TPT, as per standard of care.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis acquisition following exposure is a common occurrence, but it remains challenging to diagnose, often requiring serial testing, as immunological responses (e.g., tuberculin skin test or interferon-gamma release assays) can take weeks to provide evidence of infection. Although tuberculosis infection is generally asymptomatic, research has shown that active mycobacterial replication and inflammation occur, and its long-term effects are not well understood due to the complexity of host-pathogen interactions and delayed disease progression. While antituberculosis prophylaxis has traditionally aimed at preventing the progression from established tuberculosis infection to active tuberculosis disease, recent studies suggest that prophylaxis administered during the "window period" after exposure may also prevent its acquisition, particularly in very young children.

This trial will help determine the effectiveness of tuberculosis prophylaxis administered during the window period in preventing the acquisition of tuberculosis infection in children and adolescents exposed in household settings. If successful, the findings may inform broader strategies for tuberculosis prevention, particularly in reducing reservoirs of Mycobacterium tuberculosis and contributing to the global tuberculosis elimination efforts.

ELIGIBILITY:
Inclusion Criteria:

* Household contacts of patient (index case) with a new diagnosis of microbiologically confirmed pulmonary tuberculosis
* Age ≥5 to <18 years old

Exclusion Criteria:

* Suspected active tuberculosis in initial assessment (clinical or radiological)
* Current pregnancy or breastfeeding
* Immunocompromised
* Allergy or contraindication to isoniazid or rifapentine
* Chronic liver disease or alcohol use disorder
* History of previous treatment for active or latent tuberculosis infection
* Previous tuberculin skin test
* Household contacts of a tuberculosis index patient with a known or suspected drug-resistant M. tuberculosis strain
* Household contacts or a tuberculosis index patient currently living away from home for more than four weeks
* Household contacts of a tuberculosis index patient who have already received more than 15 daily doses of antituberculous treatment

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 647 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of new tuberculosis infections (all IGRA conversions) from enrollment until the end of follow-up in both study arms | At the end of follow-up at 12 weeks (accepted range: ≥ 12 - ≤16 weeks)

SECONDARY OUTCOMES:
Incidence of new tuberculosis infections (IGRA conversions) with high IGRA thresholds (IFN-γ ≥1.0 IU/mL) at the end of follow-up in both study arms | At the end of follow-up at 12 weeks (accepted range ≥12 - ≤16 weeks)
Incidence of active tuberculosis development until the end of follow-up in both study arms | From 4 weeks after enrollment to the end of follow-up at 12 weeks (accepted range ≥ 4 - ≤16 weeks)
Prevalence of tuberculosis infections (all IGRA positive) at the end of follow-up in both study arms | At the end of follow-up at 12 weeks (accepted range ≥ 12 - ≤16 weeks)
Incidence of 3HP-related adverse events at 12 weeks in both study arms | From TPT initiation to completion or last dose received, in both study arms (accepted range ≥ 1 day - ≤16 weeks)
To evaluate temporal changes in IFN-γ levels between baseline and follow-up among individuals receiving or not receiving tuberculosis preventive treatment | At the end of follow-up at 12 weeks (accepted range: ≥ 12 - ≤16 weeks)

CONTACTS AND LOCATIONS:
Locations (13):
- Chile (13):
  - Hospital Dr. Carlos Cisterna, Calama, Antofagasta
  - Hospital de Coquimbo, Coquimbo, Coquimbo Region
  - Hospital San Juan de Dios de La Serena, La Serena, Coquimbo Region
  - Hospital Claudio Vicuña, San Antonio, Región de Valparaíso
  - Hospital Dr. Gustavo Fricke, Viña del Mar, Región de Valparaíso
  - Hospital de Niños Roberto del Río, Independencia, Santiago Metropolitan
  - Hospital Luis Calvo Mackenna, Providencia, Santiago Metropolitan
  - Complejo Asistencial Dr. Sótero Del Río, Puente Alto, Santiago Metropolitan
  - Hospital CRS El Pino, San Bernardo, Santiago Metropolitan
  - Hospital Clínico Félix Bulnes, Santiago, Santiago Metropolitan
  - Hospital Clínico San Borja Arriarán, Santiago, Santiago Metropolitan
  - Hospital San Juan de Dios de Santiago, Santiago, Santiago Metropolitan
  - Hospital Alto Hospicio, Alto Hospicio, Tarapacá

IPD SHARING:
Plan to Share IPD: Undecided